CLINICAL TRIAL: NCT04119193
Title: Agreement and Precision of a Novel Smartphone Application (OPTIBP) For Continuous Blood Pressure Monitoring: A Comparison With the Invasive Radial Arterial Catheter
Brief Title: Agreement and Precision of a Smartphone Application For Continuous Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Other Study IDs: 2019-375
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Technology
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Novel smartphone application for blood pressure measurement — Continuous blood pressure measurements will be compared between the new application and the reference method (invasive radial arterial line) during 5 minutes of recordings.

SUMMARY:
Evaluation of an novel smartphone algorithm designed to estimate blood pressure based on collected optical signals on patients against the reference method, (radial arterial catheter) in patients admitted in the post anesthesia care unit after major surgeries.

DETAILED DESCRIPTION:
The purpose of the study is to compare the blood pressure values measured by a mobile application used with a smartphone and the values measured by reference method, which is the radial arterial line

Patients admitted to the post-anesthesia care unit after major surgeries (Erasme hospital)

Patient's arterial pressure will be measured with both measurement methods (novel smartphone application and the invasive arterial line).

The placement of an arterial line is standard of care in the investigators institution for patients scheduled for major surgeries. These patients spend 24 hours in the post-anesthesia care unit after their surgery for acute care management. Patient's blood pressure will be measured in parallel (same arm) with the mobile application and with the reference equipment (radial arterial line). Measures will be done during five times ( so five times one minute of recordings).

Blood pressure values obtained by the two methods will be compared to confirm the reliability of the data obtained with the mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in the post-anesthesia care unit after major surgery
* equipped with an arterial catheters for perioperative management
* Informed Consent as documented by signature
* Good understanding of written and oral speaking

Exclusion Criteria:

* Patients that cannot sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation
* Known contact dermatitis to nickel/chromium
* Dyshythmia like bigeminy, trigeminy, isolated Ventricular Premature Beats (VPB), atrial fibrillation
* Lesion or deficiency on hand, preventing index obstruction of smartphone's camera

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients in the post-anesthesia care unit after their major surgery, equipped with an arterial line
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Comparison of blood pressure measurement done with the novel smartphone application versus the reference method | Day of surgery
  Comparison of values to invasive reference method (arterial line)

SECONDARY OUTCOMES:
Number of necessary measure to have a good relationship between both methods | Day of surgery
  Number of necessary measure to have a good relationship between both methods
Usability assessment | Day of surgery
  Identification of possible use error in the manipulation of the device and in the performance of the measure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre J Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No